CLINICAL TRIAL: NCT00216242
Title: A Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy of Fluviral™ Influenza Vaccine in Healthy Adults 18 to 49 Years of Age
Brief Title: Study of the Protective Effect of an Injectable Influenza Vaccine Against Influenza Illness in Adults Under 50 y.o.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ID Biomedical Corporation, Quebec (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: IDB707-106
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-12-11 (Estimated); Status verified 2006-12

CONDITIONS: Influenza
Keywords: influenza; vaccine; efficacy; safety; immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza virus vaccine (Fluviral)
Biological: Saline placebo

SUMMARY:
The goal of this study is to determine whether Fluviral, an inactivated, injectable trivalent influenza vaccine (flu shot) is effective in preventing respiratory illnesses that are severe enough to limit normal daily activities and that are shown by virus culture to be caused by influenza viruses. The study will also examine the safety of the vaccine and collect measurements of the immune system responses produced by the vaccine.

DETAILED DESCRIPTION:
Yearly influenza (flu) epidemics cause a large burden of lost work and school time among younger persons and excess hospitalizations and deaths among the elderly. Injectable flu vaccines are generally believed to be effective, but formal studies using modern culture methods to prove this are limited. This study will compare the rate of respiratory illnesses associated with positive influenza virus cultures in healthy younger adults (a group at low risk for serious influenza complications) who have received Fluviral (an injectable flu vaccine) with the rate of such illnesses in healthy younger adults who have received an injection of saline (salt water). The rate of local vaccine reactions and other symptoms will be compared between the vaccine and salt water groups, and the immune responses to the vaccine measured.

ELIGIBILITY:
Inclusion Criteria:

* Good health by history and physical exam
* Reliable access to a telephone
* Study comprehension and informed consent

Exclusion Criteria:

* Systolic BP >/= 140; diastolic BP >/= 90
* Uncontrolled medical or psychiatric illness (change in last 3 months)
* Cancer, or treatment for cancer within 3 years
* Cardio-pulmonary disease requiring chronic treatment
* Insulin dependent diabetes mellitus
* Renal dysfunction (creatinine >/= 1.7 mg/dL)
* Hemoglobinopathies
* Clotting disorders that increase the risk of IM injections
* Immunosuppressive illnesses or drugs
* History of demyelinating disease (esp. Guillian-Barre syndrome)
* Employment in professions at high risk for influenza transmission
* Household contact with high-risk individuals
* Receipt of:

  a) Immunosuppressive drugs i) systemic glucocorticoids >/= 10 mg prednisone per day ii) cytotoxic drugs b) Investigational drugs within 30 days before, or planned during, the study c) Blood products within 3 months before, or planned during, the study d) Influenza vaccine within 9 months before the study e) Other vaccines within 30 days before, or planned during, the study
* History of:

  1. Severe reactions to other influenza vaccines
  2. Allergy to egg proteins
  3. Sensitivity to mercurials
* Pregnancy/ high risk of pregnancy

  1. Positive urine pregnancy test before treatment
  2. Women of child-bearing potential without credible contraceptive plan

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7400
Dates: Start 2005-09; Study Completion 2007-05

PRIMARY OUTCOMES:
Incidence of culture confirmed influenza-like illness due to virus strains matching the vaccine during the interval from November to April following treatment.

SECONDARY OUTCOMES:
Incidence of culture and/or serologically-confirmed influenza-like illness during the interval from November to April following treatment;
Rate of solicited local and systemic common reactions in days 0 to 3 post-treatment;
Rate of other adverse events through approximately 135 days post-treatment;
Rate of four-fold rises in influenza specific antibody titers 21 days after treatment;
Rate of influenza-specific antibody titers equal to, or greater than, 40 at 21 days after treatment;
Geometric mean influenza-specific antibody titers at 21 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bouveret, MD, Study Director — ID Biomedical of Quebec
Locations (41):
- United States (41):
  - Benchmark Research, Sacramento, California
  - Benchmark Research, San Francisco, California
  - Radiant Research, Denver, Colorado
  - Longmont Med. Research Center, Longmont, Colorado
  - Miami Research Associates, Miami, Florida
  - University Clinical Research Associates, Pembroke Pines, Florida
  - Emory University, Atlanta, Georgia
  - Radiant Research, Atlanta, Georgia
  - Dwight D. Eisenhower Army Medical Center, Fort Eisenhower, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Radiant Research, Boise, Idaho
  - Radiant Research, Chicago, Illinois
  - Preventive Intervention Center, Iowa City, Iowa
  - Johnson County ClinTrials, Lenexa, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Rockville Internal Medicine Group, Rockville, Maryland
  - Meridian Clinical Research, Omaha, Nebraska
  - Anderson and Collins Clinical Research, Edison, New Jersey
  - Regional Clinical Research, Endwell, New York
  - Wake Research Associates, Raleigh, North Carolina
  - National Carolina Children and Adult Clinical Research Foundation, Sylva, North Carolina
  - Carolina medical Trials, Winston-Salem, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Omega Clinical Trials, Warwick, Rhode Island
  - Radiant Research, Anderson, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Clinical Research Associates, Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Covance, Austin, Texas
  - Allergy and Asthma Research Associates, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - Killeen Scott and White Regional Clinic, Killeen, Texas
  - Research Across America, Plano, Texas
  - Benchmark Research, San Angelo, Texas
  - J. Lewis Research, Inc., Salt Lake City, Utah
  - J. Lewis Research, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Center for Health Studies, Seattle, Washington

REFERENCES:
- [Derived] Jackson LA, Gaglani MJ, Keyserling HL, Balser J, Bouveret N, Fries L, Treanor JJ. Safety, efficacy, and immunogenicity of an inactivated influenza vaccine in healthy adults: a randomized, placebo-controlled trial over two influenza seasons. BMC Infect Dis. 2010 Mar 17;10:71. doi: 10.1186/1471-2334-10-71. PMID 20236548